CLINICAL TRIAL: NCT04263883
Title: Randomized Control Trial of Addition of 3D Posture Corrective Orthosis to A Multimodal Program of Treatment Of NSNP.
Brief Title: RCT of Addition of 3D Posture Corrective Orthosis to A Multimodal Program of Treatment Of Chronic Postural Neck Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huang Xiaolin (Other)
Responsible Party: Sponsor-Investigator, Huang Xiaolin, professor of Rehabilitation, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJ-2019..
Record Dates: First submitted 2020-01-08; First posted 2020-02-11 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (Active Comparator): Usual Care Group: Conventional treatment: moist hot pack. manual therapy, Therapeutic Exercise.Home program routine.
  Interventions: Device: Study or Experimental Group
- Study or Experimental Group (Experimental): 1. moist hot pack.
  2. manual therapy.
  3. Therapeutic Exercise.
  4. Home program routine. 5.3D PCO to make mirror image therapy (reverse posture training) during the patient walking on motorized treadmill. For 10 weeks(3Times/week for 20 minutes).
  Interventions: Device: Study or Experimental Group

INTERVENTIONS:
Device: Study or Experimental Group — 3D PCO to make mirror image therapy (reverse posture training) during the patient walking on motorized treadmill, This way of functional training will deliver via the use of the adjustable cervicothoracic orthosis during the patient walking at approximately 2-3 miles per hour on a standard, motorized treadmill. The brace will reverse the abnormal posture according to the 3D posture analysis data. To facilitate tissue remodeling by reverse posture training, this called mirror image traction.then the ambulatory exercises by using treadmill will be performed while the patient's mirror image posture will be held by the adjustable orthosis, ambulatory exercises for 20 minutes by using treadmill based on Harrison et al., approach, this program will be repeated 2-3 times /week for 10weeks.

SUMMARY:
Nonspecific neck pain (NSNP) is one of the most common musculoskeletal problems treated by orthopedic physicians and physiotherapists. NSNP has an annual incidence rate of 38 to 73% and a lifetime prevalence of approximately 48%, leading to both economic and social problems.Due to increased disability-adjusted life-years from 17 million (95% confidence interval (CI): 11.4-23.7) in 1990 to 29 million (95% CI: 19.5-40.5) in 2016, Chronic neck pain is a common musculoskeletal disorder worldwide. No specific cause for neck symptoms assigned for most patients so it described as non-specific chronic neck pain (NSNP)

DETAILED DESCRIPTION:
Although the exact relationship between posture and NSNP is unsettled, the posture of the cervical spine appears to influence dorsal neck muscle activity at rest and during movement. Additionally, the forward head posture associated with thoracic kyphosis indirectly affects cervical flexion and rotational range of motion (ROM) also sustained computer work and prolonged using smart phones often in positions that encourage a functional kyphosis, appears to modify neck posture, as well as scapular positioning and upper trapezius muscle activity. Besides that Ergonomic intervention, including adjustments of the workplace station and postural correction, have been demonstrated to be effective in reducing NP with some work conditions. In addition, modalities that used to correct sagittal alignment of the cervical spine proved statistical and clinically significant results related to pain, disability, and improved nerve function. That is accomplish cause and effect relationship between bad posture and neck symptoms. According to the systematic review of Anabela et al., about head posture assessment useful for neck patients or not? The answer, of course, was yes, but it must be considered in relation to the patient's symptoms and related functional problems. Harrison and his colleagues reported that posture abnormalities occurred in the head, ribs, and pelvis in three dimensions in the form of translations and rotational displacements. Therefore, we should consider three dimensional (3D)postural assessment and correction during the treatment of NSNP associated with significant posture problems of the head in relation to thoracic. Growing research about using mirror image traction during ambulatory exercise, which is prescribed specifically to help normalize the patient's neuromuscular dysfunction and postural deformation via reflecting the patient's posture across different planes, is more beneficial than a less personalized program. With these considerations in mind and to combine the findings of 3D postural assessment into the treatment program, we designed adjustable 3D posture corrective orthotic (PCO) to be worn by the patient for a short time. The device has the ability to reflect all transitional displacements and rotational movements of the head then ask the patient to make ambulatory exercise using a treadmill while the PCO holds the patient's reverse posture. To our knowledge, no randomized clinical trial (RCT) had evaluated the addition of a 3D adjustable PCO to usual care program and investigate its short- and moderate-term improvement effects on NSNP management outcomes (i.e., neck pain, neck disability and 3-dimensional posture parameters of the head). The primary aim of our study was to evaluate of conducting an RCT using neck disability index (NDI )and 3D posture parameters. The secondary aim was NPRS and Active CervicalROM. investigate the effect size of the addition of ambulatory mirror-image traction via the wearing of 3D adjustable PCO compared to control group interventions for neck pain, disability, and 3D posture parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with age from 17-40 years old.
* Neck pain with equal or greater than 3/10 on a The Numeric Pain Rating Scale (NPRS) and the pain lasted more than 3 months (chronic neck pain).
* Participants with neck disability at least score on neck disability index (NDI) was 5 from the total score 50.
* Participants were included if they had posture deviations by screening test using GPS
* Posture displacements:

  1. An anterior head translation more than 2.5 cm.
  2. Side shifting of the head in related to thoracic more than .5 cm.

Posture rotations:

1. Rotation of head more than or equal three degrees.
2. Side bending of the head more than or equal three degrees.
3. Flexion or extension position of the head, normal angle 18 degrees, if more than that degree, it is meaning extension in upper cervical and if less means flexion in upper cervical. Participants included if they had at least two posture deviations whatever displacements or rotations. We included more obvious degrees or displacement of head posture related to thoracic to avoid variability of measurement between people and the posture deviations could be appeared and examined by visual examination.

   * If subjects could be able to continue treatment for 10 weeks then for 3 months of follow up.
   * If Participants accepted and signed an informed consent form.

Exclusion Criteria:

• If Participant reported any of the following conditions: Neck pain associated with whiplash injuries, medical red flag history(such as a tumor, fracture, metabolic diseases, rheumatoid arthritis, and osteoporosis).

* Neck pain with cervical radiculopathy, neck pain associated with externalized cervical disc herniation.
* Fibromyalgia syndrome, to avoid the similarity of fibromyalgia with an NP diagnosis, a physician used the criteria for the clinical diagnosis of fibromyalgia according to the American College of Rheumatology.
* If the patient made surgery in the neck area before whatever the cause of operation.
* Neck pain accompanied by vertigo caused by vertebrobasilar insufficiency or accompanied by non-cervicogenic headaches.
* People were excluded if they were undergoing any type of pain treatment they have psychiatric disorders or other problems that contraindicate the use of the techniques in this study.
* If Participants reported any of the following conditions: (1) a history of cervical or facial trauma or surgery. (2) Congenital anomalies involving the spine (cervical, thoracic, lumbar). (3) Bony abnormalities such as scoliosis.(4) Any systemic arthritis. (5) Recurrent middle ear infections over the last5 years or any hearing impairment requiring the use of a hearing aid. (6)Persistent respiratory difficulties over the last 5 years that had necessitated absence from work, required long-term medication or interfered with daily activities. (7) Any visual impairment not corrected by glasses. (8) Any disorder of the central nervous system. (9) pregnancy or breastfeeding because these conditions affect head posture.
* Participants could be unable to attend a 10-week treatment program and follow-up as¬sessments after 3 months.

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index, assessing change of disability of neck patients | Pre treatment at 1st day , post treatment after 10 weeks , follow up after 6 months.
  The NDI is a modification of the Oswestry Low Back Pain Disability Index. It is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. The NDI has sufficient support and usefulness to retain its current status as the most commonly used self-report measure for neck pain The NDI can be scored as a raw score [2]or doubled and expressed as a percent [3]. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means worst imaginable pain'. All the points can be summed to a total score. The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage.0 points or 0% means no activity limitations, 50 points or 100% means complete activity limitation.
Three-dimensional posture parameters of the head in relation to thoracic measured by global posture system (GPS) device.assessing the change of posture of neck patients | Pre treatment at 1st day , post treatment after 10 weeks , follow up after 6 months.
  Postural translation of the head
  1. Tx(mediolateral translation )
  2. Tz(anteroposterior translation ) Postural rotations of the head
  1.Rx(flexion or extension position) 2.Ry (r.t rot. or l.t rot.) 3.Rz (r.t side bending or l.t side bending)

SECONDARY OUTCOMES:
The Numeric Pain Rating Scale (NPRS) | Pre treatment at 1st day , post treatment after 10 weeks , follow up after 6 months.
  is an 11-point numeric pain intensity ranging from 0 ('no pain') to 10 ('as much pain as possible'). A change of two points or more was identified as the minimal clinically important difference in patients with chronic neck pain.
Active cervical ROM using CROM | Pre treatment at 1st day , post treatment after 10 weeks , follow up after 6 months.
  with an inclinometer (CROM Deluxe model, Performance Attainment Associates, Lindstrom, Minnesota).The CROM consists of 2 gravity-dependent goniometers, one compass dial, and a head-mounted frame allowing measurement of ROM in 3 planes (flexion/ extension, lateral flexion, rotation). A magnetic yoke consisting of 2 bar magnets held anteriorly and posteriorly was provided to reduce the influence of thoracic rotation. The CROM has demonstrated good concurrent validity for active ROM. According to the systematic review by Chen et al, the mean normative values of cervical ROM were determined to be: 52 degrees for flexion, 71 degrees for the extension, 72degrees for rotation, and 43 degrees for lateral flexion. Documentation of cervical ROM was rendered in the form of the full range (ie, a total value for the sagittal, frontal, or transverse plane, yielding 3 measurements).
Zung Self-Rating Anxiety Scale (SAS) | Pre treatment at 1st day , post treatment after 10 weeks , follow up after 6 months.
  The SAS test is self-administered, with each response using a 4-point scale, from 'none of the time" to "most of the time." There are 20 questions with 15 increasing anxiety level questions and 5 decreasing anxiety questions. There are two formats, self-evaluations, and clinical evaluations.
Tampa Scale of Kinesiophobia (TSK) | Pre treatment at 1st day , post treatment after 10 weeks , follow up after 6 months.
  Kinesiophobia was assessed with the 13-item Chinese version of the Tampa Scale of Kinesiophobia (TSK)

OTHER OUTCOMES:
Global Perceived Effect Questionnaire (GPE) | post treatment after 10 weeks , follow up after 6 months.
  The perceived effect of the intervention was assessed with the Global Perceived Effect Questionnaire. 5-point Likert-type scale used to evaluate self-reported improvement or deterioration after the intervention. The use of the GPE is widely reported in the physical therapy literature. Patient satisfaction was assessed with the Chinese version of the PhysicalTherapy Patient Satisfaction Questionnaire (PTPSQ-I[ which demonstrated good psychometric properties and a 2-factor structure, related to perceived "overall experience" and "professional impression." (GPE),

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin Huang, Professor, Study Director — Tongji Hospital
Locations (1):
- TongjiHospital, Wuhan, Hubei, China